CLINICAL TRIAL: NCT01740089
Title: Multicenter Open-label Randomized Prospective Clinical Study of Efficacy and Safety of Algeron (Cepeginterferon Alfa-2b) in Comparison With PegIntron (Peginterferon Alfa-2b) in the Combined Treatment of Chronic Hepatitis C
Brief Title: Algeron (Cepeginterferon Alfa-2b) Compared With PegIntron (Peginterferon Alfa-2b) for Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG-IFNа-2
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis; Hepatitis C
Keywords: Hepatitis C; Cepeginterferon alfa; Peginterferon; Treatment
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Algeron 1.5 μg/kg (Experimental): Algeron 1.5 μg/kg of body weight weekly subcutaneously in combination with ribavirin daily orally in a daily dose of 800 mg (patients with body weight < 65 kg), 1000 mg (patients with body weight of 65-85 kg inclusive), 1200 mg (patients with body weight of 86-105 kg inclusive) or 1400 mg (patients with body weight > 105 kg).
  Interventions: Drug: Algeron; Drug: Ribavirin
- Algeron 2.0 μg/kg (Experimental): Algeron 2.0 μg/kg of body weight weekly subcutaneously in combination with ribavirin daily orally in a daily dose of 800 mg (patients with body weight < 65 kg), 1000 mg (patients with body weight of 65-85 kg inclusive), 1200 mg (patients with body weight of 86-105 kg inclusive) or 1400 mg (patients with body weight > 105 kg).
  Interventions: Drug: Algeron; Drug: Ribavirin
- PegIntron (Active Comparator): PegIntron 1.5 μg/kg of body weight weekly subcutaneously in combination with ribavirin daily orally in a daily dose of 800 mg (patients with body weight < 65 kg), 1000 mg (patients with body weight of 65-85 kg inclusive), 1200 mg (patients with body weight of 86-105 kg inclusive) or 1400 mg (patients with body weight > 105 kg).
  Interventions: Drug: PegIntron; Drug: Ribavirin

INTERVENTIONS:
Drug: Algeron — 1.5 μg/kg or 2.0 μg/kg of body weight weekly subcutaneously
  Other Names: cepeginterferon alfa-2b
  Arms: Algeron 1.5 μg/kg; Algeron 2.0 μg/kg
Drug: PegIntron — 1.5 μg/kg/week subcutaneously in combination with ribavirin
  Other Names: Peginterferon alfa-2b
  Arms: PegIntron
Drug: Ribavirin — 800-1400 mg/day orally

SUMMARY:
The purpose of the study is to demonstrate the noninferiority of Algeron 1.5 and 2.0 μg/kg/week in combination with ribavirin compared to PegIntron in combination with ribavirin in the treatment of chronic hepatitis C, and to determine therapeutic dose of Algeron.

DETAILED DESCRIPTION:
After 12 weeks of treatment, an assessment of treatment efficacy was performed, i.e. rates of rapid (after 4 weeks) and early (after 12 weeks) virologic responses according to serum HCV RNA level PCR data. In patients without virologic response after 12 weeks, AVT was discontinued, and they were withdrawn from the study. Patients with EVR were enrolled in a follow-up period. During the follow-up period, patients of the first and the second group will receive Algeron in the selected therapeutic dose in combination with ribavirin, patients of the third group - PegIntron in combination with ribavirin during 12 or 36 weeks (depending on a genotype of the virus), afterwards they will be followed up without therapy for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Hepatitis С virus infection (genotypes 1а, 1b, 2, 3, 4) confirmed by a positive quantitative PCR (HCV RNA > 50 IU/ml).
3. Males and females aged from 18 to 70 years inclusive.
4. Body mass index of 18 - 30 kg/m inclusive.
5. Increased ALT level (> 40, < 400 IU/L), documented at least twice within the last 6 months.
6. Preserved protein synthetic liver function (i.e. INR < 1.7, albumin > 35 g/l).
7. No signs of hepatic encephalopathy or abdominal fluid retention according to clinical and ultrasound examination.
8. Fertile patients and their partners agree to use barrier contraception throughout the study and 7 months after its completion.

Exclusion Criteria:

1. Intolerance of IFN alpha formulations, ribavirin or any components of these drugs according to the past medical history.
2. Infection by hepatitis B virus or HIV.
3. Past history of HCV treatment with IFN alfa or pegylated IFN alfa formulations.
4. Administration of interferons and/or interferon inducing drugs for any indication within 1 month prior to the enrollment into the study.
5. Cholestatic hepatitis (conjugated bilirubin, alkaline phosphatase, ALT levels of more than 5 ULN).
6. Decompensated liver cirrhosis confirmed by laboratory findings (Child-Pugh class B, С) or ultrasound examination.
7. Any documented autoimmune diseases.
8. Hematologic (hemoglobin < 130 g/L for males and < 120 g/L for females; neutrophils < 1.5 х109/L; platelets < 90 х109/L) or biochemical abnormalities (creatinine level of more than 1.5 ULN, creatinine clearance less than 50 mL/min).
9. Documented diagnosis of hemoglobinopathies (e.g., thalassemia major, sickle-cell anemia).
10. Heavy depression, any other mental disorders, which in the Investigator's opinion can be contraindications for antiviral treatment.
11. Epilepsy and/or other functional disorders of the central nervous system.
12. Abnormal thyroid function (TTH level beyond the normal values).
13. Malignant neoplasms.
14. Pregnancy, lactation period.
15. Severe comorbidities (for example, severe hypertension, severe coronary heart disease, decompensated diabetes mellitus), which in the Investigator's opinion can be contraindications for antiviral treatment.
16. Documented rare hereditary diseases, such as intolerance of lactose, sucrose, fructose, lactase deficiency or glucose-galactose malabsorption.
17. Current alcohol or drug abuse, which in the Investigator's opinion can be contraindications for antiviral treatment or restrict treatment compliance.
18. Simultaneous participation in other clinical trials or prior participation in this or another clinical trial within less than 30 days after its completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Znoyko, professor, Principal Investigator — Moscow State University of Medicine and Dentistry; Marina Maevskaya, professor, Principal Investigator — The First Moscow State Sechenov Medical University; Svetlana Kizhlo, Principal Investigator — Health Department "Center for Prevention and Control of AIDS and Infectious Diseases"; Natalia Petrochenkova, Principal Investigator — Smolensk State Medical Academy; Semen Maximov, Principal Investigator — Moscow State University of Medicine and Dentistry; Firaja Nagimova, Principal Investigator — Kazan State Medical University; Vladimur Yakovlev, Principal Investigator — 7. St. Petersburg State Institution of Health "Clinical Infectious Diseases Hospital named SP Botkin"
Locations (1):
- Moscow State University of Medicine and Dentistry, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: First 12 Weeks of Treatment
Arm/Group | Algeron 1.5 μg/kg | Algeron 2.0 μg/kg | PegIntron
Started | 50 | 50 | 50
Completed | 50 | 48 (Withdrawn due to: AE before W12 (n=1) Withdrew consent before W12 (n=1)) | 48 (Withdrawn due to: AE before W12 (n=2))
Not Completed | 0 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: After 12 Weeks
Arm/Group | Algeron 1.5 μg/kg | Algeron 2.0 μg/kg | PegIntron
Started | 50 | 48 | 48
Completed | 43 (Withdrawn due to: No EVR (n=3) AE (n=2) No EOT (n=1) Non-compliance (n=1)) | 45 (Withdrawn due to: Withdrawn consent (n=1) No EVR (n=1) Non-compliance (n=1)) | 37 (Withdrawn due to: No EVR (n=4) AE (n=5) Non-attendance of visit (n=1) Withdrawn consent (n=1))
Not Completed | 7 | 3 | 11
Not completed — Lack of Efficacy | 3 | 1 | 4
Not completed — Adverse Event | 2 | 0 | 5
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: During randomization, patients were stratified by gender, age, viral load, and HCV genotype. The mITT-analysis included all randomized patients received at least one dose of investigational products, who were not withdrawn from the study at its beginning due to serious violations of the inclusion/non-inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Algeron 1.5 μg/kg | Algeron 2.0 μg/kg | PegIntron | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [30 to 39] | 34 [29 to 42] | 36 [30 to 41] | 35 [30 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 15 | 44
  Male | 37 | 34 | 35 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 50 | 49 | 50 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 50 | 50 | 50 | 150
HCV genotype [Number; unit: participants]
  HCV 1b | 22 | 26 | 26 | 74
  HCV 1a | 4 | 1 | 2 | 7
  HCV 2 | 2 | 2 | 1 | 5
  HCV 3 | 22 | 21 | 21 | 64
Initial Viral load [Number; unit: participants]
  High (>8х10^5 IU/ml) | 17 | 16 | 14 | 47
  Low (≤8х10^5 IU/ml) | 33 | 34 | 36 | 103
Interleukin 28B (IL-28B) genotype [Number; unit: participants]
  C/C | 19 | 17 | 13 | 49
  C/T | 24 | 26 | 26 | 76
  T/T | 7 | 7 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Randomized Patients Achieving Early Virologic Response (EVR) - Negative PCR Result for HCV RNA (< 15 IU/ml) or ≥ 2log10 Decrease of Viral Load After 12 Weeks of Study Treatment.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Algeron 1.5 μg/kg | Algeron 2.0 μg/kg | PegIntron
Number analyzed (Participants) | 50 | 50 | 50
participants | 47 | 47 | 44

2. Secondary Outcome: Number of Randomized Patients Achieving Rapid Virologic Response (RVR) - Negative PCR Result for HCV RNA (< 15 IU/ml) After 4 Weeks of Treatment.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Algeron 1.5 μg/kg | Algeron 2.0 μg/kg | PegIntron
Number analyzed (Participants) | 50 | 50 | 50
participants | 32 | 28 | 33

3. Secondary Outcome: Number of Randomized Patients Achieving Sustained Virologic Response (SVR) - Negative PCR Result for HCV RNA (< 15 IU/ml) 24 Weeks After Last Dose of Study Treatment.
Time Frame: 24 weeks after last dose of study treatment
Measure: Number; unit: participants
Groups:
- Algeron (n=100): the comparative inter-group analysis of efficacy was performed for patients of groups 1 and 2 received Algeron (n=100), because after 12 weeks of therapy and analysis of data, all patients of the first and second groups continued receive Algeron in a chosen therapeutic dose 1.5 µg/kg.
Arm/Group | Algeron (n=100) | PegIntron (n=50)
Number analyzed (Participants) | 100 | 50
participants | 75 | 34

4. Secondary Outcome: Number of Patients Who Have Undetectable HCV RNA (< 15 IU/ml) at the End of Treatment.
Time Frame: After 24 weeks of treatment for patients with genotype 2 or 3 and after 48 weeks of treatment for patients with genotype 1 or 4.
Measure: Number; unit: participants
Arm/Group | Algeron (n=100) | PegIntron (n=50)
Number analyzed (Participants) | 100 | 50
participants | 88 | 38

5. Other Pre Specified Outcome: Immunogenicity
Description: Number of randomized patients with neutralizing antibodies to IFN alfa on weeks 0, 12, 24, 48 (for patients with genotype 1 or 4) and 24 weeks after last dose of study treatment.
Time Frame: Weeks 0, 12, 24, 48 (for patients with genotype 1 or 4) and 24 weeks after last dose of study treatment
Measure: Number; unit: participants
Arm/Group | Algeron (n=100) | PegIntron (n=50)
Number analyzed (Participants) | 100 | 50
participants | 0 | 0

ADVERSE EVENTS:
Description: The number of patients for the efficacy analysis was 150. 151 patients were included in the safety analysis, including 1 patient in Algeron group withdrawn at early stages due to a violation of inclusion/non-inclusion criteria [severe depression at Visit 1], who was not considered to be enrolled in the study due to serious protocol violation.
Groups:
- Algeron (n=101): The safety analysis included 101 patients received at least 1 dose of Algeron (taking into account one patient withdrawn at early stages of the study due to a protocol violation [severe depression by the Beck's scale before the first injection], who was withdrawn from the mITT-analysis)
Arm/Group | Algeron (n=101) | PegIntron (n=50)
Serious Adverse Events (participants affected / at risk) | 2/101 | 2/50
Other Adverse Events (participants affected / at risk) | 101/101 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Algeron (n=101) (N=101) | PegIntron (n=50) (N=50)
dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
drug-induced pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
phlegmonous appendicitis (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Algeron (n=101) (N=101) | PegIntron (n=50) (N=50)
Flu-like syndrome (General disorders) | 86 (86) | 49 (49)
Asthenia (weakness, fatigue) (General disorders) | 63 (63) | 22 (22)
Grade I decreased body weight (General disorders) | 25 (25) | 12 (12)
Grade II decreased body weight (General disorders) | 11 (11) | 8 (8)
Headache (Nervous system disorders) | 52 (52) | 32 (32)
Dizziness (Nervous system disorders) | 12 (12) | 5 (5)
Depression (Psychiatric disorders) | 13 (13) | 3 (3)
Irritability, emotional lability (Psychiatric disorders) | 15 (15) | 4 (4)
Sleep disorders (Psychiatric disorders) | 9 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 14 (14) | 7 (7)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 9 (9) | 3 (3)
Decreased appetite (Gastrointestinal disorders) | 10 (10) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 17 (17) | 4 (4)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 5 (5)
Dyspnoe (including dyspnoe after exercises) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 30 (30) | 24 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (33) | 16 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 27 (27) | 12 (12)
Skin itch (Skin and subcutaneous tissue disorders) | 21 (21) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 14 (14) | 6 (6)
Skin dryness and exfoliation (Skin and subcutaneous tissue disorders) | 23 (23) | 7 (7)
Stomatitis and gingivitis (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Blepharitis and conjunctivitis (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Rhinitis, nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Hoarseness, throat irritation, sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Grade 1 leucopenia (Blood and lymphatic system disorders) | 29 (29) | 13 (13)
Grade 2 leucopenia (Blood and lymphatic system disorders) | 45 (45) | 23 (23)
Grade 3 leucopenia (Blood and lymphatic system disorders) | 20 (20) | 11 (11)
Grade 1 neutropenia (Blood and lymphatic system disorders) | 11 (11) | 10 (10)
Grade 2 neutropenia (Blood and lymphatic system disorders) | 36 (36) | 14 (14)
Grade 3 neutropenia (Blood and lymphatic system disorders) | 29 (29) | 13 (13)
Grade 4 neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Grade 1 lymphopenia (Blood and lymphatic system disorders) | 8 (8) | 9 (9)
Grade 1 thrombocytopenia (Blood and lymphatic system disorders) | 47 (47) | 23 (23)
Grade 2 thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Grade 1 anemia (Blood and lymphatic system disorders) | 73 (73) | 33 (33)
Grade 2 anemia (Blood and lymphatic system disorders) | 12 (12) | 8 (8)
Increased TTH level (Endocrine disorders) | 12 (12) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No